CLINICAL TRIAL: NCT04704999
Title: Optimizing the Dose of Tafenoquine for the Radical Cure of Plasmodium Vivax Malaria in Southeast Asia
Brief Title: Southeast Asia Dose Optimization of Tafenoquine
Acronym: SEADOT
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MAL20005; 21-0023 (Other Grant/Funding Number: DMID reference)
Record Dates: First submitted 2021-01-05; First posted 2021-01-12 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-02

CONDITIONS: Plasmodium Vivax Malaria
Keywords: Plasmodium vivax; Relapse; 8-aminoquinoline; Tafenoquine; Radical cure; Drug efficacy; Adults; Pediatrics
MeSH Terms: conditions — Malaria, Vivax; Recurrence | interventions — tafenoquine; Chloroquine; Artemether; Lumefantrine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single (Outcomes Assessor) This is a double-blind randomized superiority trial. The laboratory staff responsible for reading the malaria blood smear slides will be blinded to treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tafenoquine standard dose (TQ-current) (Active Comparator): Arm 1
  * >10 kg to ≤20 kg 100 mg
  * >20 kg kg ≤35 kg 200 mg
  * >35 kg 300 mg
  Tafenoquine will be given as 100 mg coated tablets. Tablets will be given, and dosing will be based on weight bands.
  Interventions: Drug: Tafenoquine; Drug: Chloroquine; Drug: Artemether 20 mg-Lumefantrine 120 mg
- Tafenoquine 50% higher dose (TQ-higher) (Active Comparator): Arm 2
  * >10 kg to ≤20 kg 150 mg
  * >20 kg kg ≤35 kg 300 mg
  * >35 kg 450 mg
  Tafenoquine will be given as 100 mg coated tablets. Whole tablets will be given, and dosing will be based on weight bands.
  Interventions: Drug: Tafenoquine; Drug: Chloroquine; Drug: Artemether 20 mg-Lumefantrine 120 mg

INTERVENTIONS:
Drug: Tafenoquine — Tafenoquine will be given as 100mg coated tablets. Tablets will be given based on weight bands.
Drug: Chloroquine — Chloroquine will be given as daily dose over 3 days (25mg/kg total dose divided 10/10/5mg/kg)
Drug: Artemether 20 mg-Lumefantrine 120 mg — Artemether-lumefantrine will be given twice daily over 3 days. Whole tablets will be given based on weight bands.

SUMMARY:
Tafenoquine was recently approved by regulatory authorities in the USA and Australia. Tafenoquine is an alternative radical curative treatment to primaquine acting against the dormant liver stage of Plasmodium vivax (the hypnozoite). Tafenoquine (an 8-aminoquinoline) has the substantial advantage of single dosing as compared to a 14-day course of primaquine to achieve radical cure. The recommended tafenoquine dose is 300 mg, which was shown to be significantly worse in radical curative efficacy to a total primaquine dose of 3.5 mg/kg in Southeast Asia. The cure rate of tafenoquine 300 mg in Southeast Asian study sites was only 74%. The comparator 3.5 mg/kg total primaquine dose is the standard and most commonly used dose globally, but in Southeast Asia and the Western Pacific, higher doses of primaquine are needed for radical cure. This study aims to determine the optimal dose of tafenoquine in Southeast Asia.

DETAILED DESCRIPTION:
Study design

A total of 700 participants will be enrolled and randomized to one of two arms: the currently recommended tafenoquine dose (TQ-current; e.g., 300mg adult dose) or a 50% higher tafenoquine dose (TQ-higher; e.g., 450mg adult dose). Doses will be equal to 100, 150, 200, 300, or 450 mg, given as a single dose. Each arm will have 350 participants. The schizonticidal agent used will be determined by the study site. Tafenoquine will be given concomitantly with the schizonticidal agent on the day of enrolment. The participant will follow up daily until the malaria smear is negative for asexual parasites or until the schizonticidal treatment is completed, whichever occurs last. Follow up will continue on days 7, 14, 21, and 28 then every month until month 4. Participants will be instructed to follow up in between visits if they are feeling unwell. Treatment allocation will be double-blind.

Recruitment

Potential participants will be recruited from the outpatient setting at the following sites:

* Mahidol Oxford Tropical Medicine Research Unit, Cambodia
* Lao Oxford Mahosot Hospital Wellcome Trust Research Unit, Lao PDR
* Mahidol Vivax Research Unit, Thailand
* Shoklo Malaria Research Unit, Thailand
* Oxford University Clinical Research Unit, Vietnam

Screening and Enrolment

Patients presenting with fever or history of fever and have asexual P. vivax parasitemia by microscopy will be approached for informed consent. After written informed consent has been provided, study staff who have been trained in phlebotomy will draw approximately 7.14 mL of blood. Medical history, participant weight, vital signs and physical examination, point of care hemoglobin, quantitative glucose-6-phosphate dehydrogenase testing, and urine pregnancy testing will be performed for eligibility assessment.

Randomization

Randomization will be done by sequentially numbered sealed opaque envelopes and prepared by a Clinical Trials Support Group (CTSG) that is not involved with study activities. The CTSG will maintain a log of the study group allocation and control access to the log. The randomized arms will be TQ- current (the currently recommended tafenoquine dose) and TQ-higher (a 50% higher tafenoquine dose than currently recommended). Tafenoquine treatment will be double blinded so all participants will take a study drug with or without matching placebo. Participants will receive a fixed mg dose depending on their weight. The weight bands will be provided in a dosing table. Randomization will be stratified by site.

Direct Observation of Drug Administration

To ensure complete adherence to the prescribed drug regimens, all drug administration will be directly observed by study staff.

The following procedures are to be performed for each drug administration:

* Record adverse events as reported by participant or observed by study staff
* Record vital signs
* Record the date and time of study drug administration

Study staff will review any available laboratory findings prior to drug administration. The investigator will determine if any adverse event requires discontinuation of the study medication or inability to continue with study procedures.

Follow-up Visits

Participants will be followed daily until the malaria smear is negative once or when the schizonticidal treatment is completed, whichever is later. Follow up will continue on days 7, 14, 21, and 28, then months 2, 3, and 4 (total of 10 visits depending on parasite clearance time). Daily visits must occur on the exact day scheduled. The visit windows for the day 7, 14, and 21 visits are +/- 3 days, for the day 28 visit + 2 weeks/- 3 days, and for the months 2, 3, and 4 visits are +/- 2 weeks. The following procedures are to be performed for each visit:

* Medication history and concomitant medication use
* Record adverse events as reported by participant or observed by study staff
* Record vital signs and physical examination
* Collect blood samples for laboratory tests
* Review all available laboratory results

At study exit on month 4, any participant with ongoing, unresolved adverse events will be referred for appropriate outpatient clinical follow-up. If the participant has a P. vivax recurrence, they will be treated as per the randomization arm and study activities (blood sampling and follow up) will restart as episode 2, day 0. The total study duration will remain the same. This means that the study completion date is 4 months from the date of enrolment for all participants regardless of the number of P. vivax episodes.

Missed Visits

If the participant does not show for a scheduled study visit, study personnel will call the participant or visit their home to remind the participant of the study visit. Maximum efforts will be made to ensure complete follow-up in the trial, including routine education for participants on follow up schedules. If the scheduled visit is not completed within the window period, that visit will be documented as "missed" and follow up will continue.

Participant Withdrawal or Termination

Each participant has the right to withdraw consent for the study at any time. In addition, the investigator may discontinue a participant from the study at any time if the investigator considers it necessary for any reason including:

* Ineligibility (arising during the study or retrospective having been overlooked at screening)
* Significant non-compliance with treatment regimen or study requirements
* An adverse event which requires discontinuation of the study medication or results in inability to continue to comply with study procedures

The reason for withdrawal will be recorded in the case report form (CRF). If the participant is withdrawn due to an adverse event, the investigator will arrange for follow-up visits or telephone calls until the adverse event has resolved or stabilized. Participants who have been withdrawn or terminated from the study will not be replaced.

Sample Size

The trial hypothesis is that the radical cure efficacy of TQ-higher is at least 10% greater than TQ-current. This will be assessed by the absence of recurrent P. vivax infection by 4 months. From previous data in the pre-registration trials, TQ-current had a radical cure efficacy of approximately 74% by 6 months. In short latency settings, over 90-95% of the recurrences occur within 4 months thus, the 4-month endpoint should have a high sensitivity. To detect a 10% difference between TQ-current and TQ-higher, account for 25% loss to follow up, and achieve at least 80% power a sample size of about 350 participants in each arm is needed. The sample size calculation as done in Stata 17 using the following command "power twoproportions 0.74, diff(0.10)" and was then adjusted for a 25% loss to follow-up. Significance level (alpha) will be set at 0.05 using a two-sided two-sample proportions z-test. Therefore, a total of 700 participants will be enrolled across 5 countries (~140 participants in each country). Enrolment may be shifted to other countries if recruitment rates in a country do not meet study timelines.

DATA HANDLING AND RECORD KEEPING

Data Collection

All study data will be recorded on standard paper Case Report Forms (CRFs). Data will be entered on a secure database in accordance with standard operating procedures (SOPs). A study-specific data management plan will detail procedures for collection, curation, and storage of study data. For most variables, the CRF will be considered the source document.

All documents will be stored safely in confidential conditions. On all study specific documents, other than the signed consent and screening logbook, the participant will be referred to by the study participant number/code, not by name.

Data Access

The participants will be identified by a study identification number in the study database. The name and any other identifying detail will NOT be included in any study data electronic file. The database linking the volunteer's clinical identification number (ie. hospital number) to the study identification number will be kept by the individual study sites and the data analysis team will not have access to this information. All records will be kept locked and all databases will be password protected and only clinic staff and study staff will have access to their respective databases. Direct access will be granted to authorized representatives from the sponsor, host institutions and the regulatory authorities to permit trial-related monitoring, audits and inspections.

Data Storage

Each study site will maintain, and store securely, complete, accurate and current study records throughout the study. In accordance with the University of Oxford's policy, research data and records should be retained for five years for adults, and for children until the youngest child participating in the trial reaches 21, or in accordance with the local/in-country regulation. Applicable records include source documents, site registration documents and reports, informed consent forms, and notations of all contacts with participants.

Data Sharing

Participant's data and results from blood analyses stored in the database may be shared according to the terms defined in the MORU data sharing policy or other researchers to use in the future. All personal information will be anonymized so that no individual can be identified from their treatment records.

Quality Control and Quality Assurance

The study will be conducted with the current approved protocol, International Conference on Harmonisation (ICH) Good Clinical Practice (GCP), relevant regulations, standard operating procedures, and the General Data Protection Regulation (GDPR). The Clinical Trials Support Group (CTSG) at MORU will provide study oversight, quality management, and study monitoring.

Statistical Analysis

Baseline participant characteristics will be described by treatment arms as either mean and standard deviation, median and interquartile range and/or full range, or expressed as frequency and percentage depending on the data characteristics. We will perform an intention-to-treat (ITT) analysis where participants will be analyzed according to the arm of randomization irrespective of the treatment that was actually given and participant adherence to the study drug. Multiple imputation (MI) will be used for handling missing outcome data each missing value having 5 multiply imputed values that will be combined using Rubin's rule [Rubin DB. 1996]. These analyses will be followed by complete case (CC) analysis. To assess the differences in the primary and secondary endpoints (microscopy and sub-microscopic P. vivax recurrence by month 4, respectively) between treatment arms, a generalized linear models for the binomial family with identity link will be used to obtain risk differences and the corresponding 95% confidence interval (CI). A multivariable mixedeffects generalized linear models for the binomial family with identity link will be fitted for the primary outcome. This model will include random intercepts for country and site, and explanatory variables such as demographic factors and baseline characteristics; the schizonticidal drug (chloroquine and artemetherlumefantrine); tafenoquine mg/kg dose, AUC, Cmax, t1/2; potential tafenoquine metabolites; CYP2D6 status, and methemoglobin level. Survival analysis will be used to evaluate time to microscopy positive P. vivax recurrence. For the adverse event analysis, Fisher's exact test will be used for binary data. Hemoglobin and methemoglobin levels and association with drug exposure will be analyzed using linear regression. The estimated tafenoquine AUC model will be based on previous work on primaquine pharmacokinetic-pharmacodynamic analysis using nonlinear mixed-effects modelling. A detailed statistical analysis plan (SAP) will be developed as a separate document and will be finalized before the database is locked and the details of analysis for the secondary outcomes will be in the SAP.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic P. vivax mono-infection as diagnosed by microscopy
* Fever or history of fever in the previous 7 days
* Quantitative G6PD activity ≥70% of the population median
* Weight >10 kg and ≥2 years old
* Ability to understand the study instructions and provide written informed consent.
* Willing to be followed for 4 months

Exclusion Criteria:

* Pregnancy
* Lactation
* Hb < 8 g/dL
* Severe malaria
* Blood transfusion in the last 4 months
* History of allergic response to an 8-aminoquinoline or the nationally recommended schizonticide (e.g., chloroquine, artemether-lumefantrine)
* Any previous history of a haemolytic event Presence of any condition which in the judgement of the investigator would place the patient at undue risk or interfere with the results of the study (e.g. chronic disease, medications that potentiate or inhibit CYP2D6 or CYP2C8 isoenzyme function)

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2024-07-22 (Actual); Primary Completion 2027-10-04 (Estimated); Study Completion 2028-02-07 (Estimated)

PRIMARY OUTCOMES:
Microscopy positive P. vivax recurrence after radical treatment up to month 4 | At month 4

SECONDARY OUTCOMES:
Sub-microscopic P. vivax recurrence after radical treatment between day 28 and month 4 | At Day 28; Month 4
Sub-microscopic P. vivax recurrence with very low parasite density after radical cure treatment at days 14 and 21 | At Day 14 and 21
Number of serious adverse events (e.g., hospitalization for symptomatic hemolysis or methemoglobinemia) | At Days 1, 2, 7, 14 and Months 1, 2, 3, 4
Number of adverse events (e.g., gastrointestinal symptoms) | At Days 1, 2, 7, 14 and Months 1, 2, 3, 4
Methemoglobin levels measured by pulse oximetry at day 7 | At Day 7
Tafenoquine AUC and t1/2 as estimated from plasma tafenoquine concentrations at days 0, 1, 2, and 7, and monthly visits until month 4 | At Day 0, 1, 2, and 7; Month 1, 2, 3, and 4
Plasma tafenoquine concentrations at days 0, 1, 2, and 7, and at monthly visits until month 4 | At Day 0, 1, 2, and 7; Month 1, 2, 3, and 4
Tafenoquine metabolites identification in red blood cell and urine at days 1, and 2 or 3 | At Day 1, 2, and 3
The probability of treatment failure defined as by the probability of one or more of the observed recurrences within 4 months being a relapse, using time-to-event and estimated identity-by-descent of recurring parasite genotypes compared to enrolment | At Day 0, 7, 14, 21, and 28; Month 2, 3, and 4

CONTACTS AND LOCATIONS:
Overall Officials: Cindy Chu, MD, PhD, Principal Investigator — Lao-Oxford-Mahosot Hospital-Wellcome Research Unit
Locations (5):
- Mahidol Oxford Tropical Medicine Research Unit (MORU), Cambodia, Siem Reap, Cambodia
- Lao Oxford Mahosot Hospital Wellcome Trust Research Unit (LOMWRU), Vientiane, Laos
- Thailand (2):
  - Mahidol Vivax Research Unit (MVRU), Bangkok
  - Shoklo Malaria Research Unit (SMRU), Bangkok
- Oxford University Clinical Research Unit (OUCRU), Bình Phước, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Participant's data and results from blood analyses stored in the database may be shared according to the terms defined in the MORU data sharing policy or other researchers to use in the future. All personal information will be anonymized so that no individual can be identified from their treatment records. The genomic data sharing plan will be shared on a public database and the plan will be kept in the Regulatory Binder (or manual of procedures).